CLINICAL TRIAL: NCT02118376
Title: Effects of GLP-1 Receptor Agonist on Fat Redistribution and Inflammatory Status in Female Patients With Type 2 Diabetes and Obesity
Brief Title: Effects of GLP-1 Receptor Agonist on Fat Redistribution and Inflammatory Status
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai 10th People's Hospital (Other)
Responsible Party: Principal Investigator, Zhang Manna, Professor, Shanghai 10th People's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GLP-1
Record Dates: First submitted 2013-12-20; First posted 2014-04-21 (Estimated); Last update posted 2014-04-21 (Estimated); Status verified 2013-12

CONDITIONS: Obesity
Keywords: obesity; fat distribution; inflammation
MeSH Terms: conditions — Obesity; Inflammation | interventions — Exenatide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- exenatide (Experimental): exenatide, 5ug, bid, 3months
  Interventions: Drug: Exenatide

INTERVENTIONS:
Drug: Exenatide — 5ug bid,Subcutaneous injection
  Other Names: Byetta

SUMMARY:
GLP-1 receptor agonists promote fat redistribution in obese women with type 2 diabetes, reduce liver fat content, improve the inflammation state

DETAILED DESCRIPTION:
As a treatment for type 2 diabetesGlucagon like peptide -1 (Glucan-like peptide-1, GLP-1) receptor agonists plays the role of promoting insulin secretion, inhibiting glucagon secretion，and also has the central and peripheral effects,it can inhibit appetite,reduce weight.GLP-1 receptor agonists promote fat redistribution in obese women with type 2 diabetes, reduce liver fat content, improve the inflammation state

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of overweight and type 2 diabetes mellitus

Exclusion Criteria:

* Poor body condition (severe liver and kidney dysfunction)
* Unknown causes of pancreatitis, chronic pancreatitis, pancreatic resection, stomach operation, malignant tumor, previous use of systemic corticosteroids (local or inhalation of exceptions) heart function or niacin, incomplete
* serious endocrine disease
* genetic disease

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2014-08; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Dual energy X-ray absorptiometry | 3 month
  fat distribution

SECONDARY OUTCOMES:
lab testing | 3 month
  inflammation

OTHER OUTCOMES:
lab testing | 3 months
  liver function

CONTACTS AND LOCATIONS:
Overall Officials: Qu Shen, Study Director — Shang Tenth People's Hospital
Locations (1):
- Shanghai Tenth People' Hospital, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Wang X, Chen J, Li L, Zhu CL, Gao J, Rampersad S, Bu L, Qu S. New association of bone morphogenetic protein 4 concentrations with fat distribution in obesity and Exenatide intervention on it. Lipids Health Dis. 2017 Apr 4;16(1):70. doi: 10.1186/s12944-017-0462-1. PMID 28376799